CLINICAL TRIAL: NCT03688022
Title: An Open Label, Multicentre, Randomised, 2-cohort, Sequential and Crossover Study to Assess the Relative Oral Bioavailability of MT-7117 Higher Content Tablets Versus MT-7117 Lower Content Tablets and the Pharmacokinetics of MT-7117 Under Various Gastric Conditions in Healthy Subjects
Brief Title: Relative Bioavailability and Drug-drug Interaction Study With MT-7117 and a Proton Pump Inhibitor
Acronym: MT-7117 BA DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MT-7117-E03; 2018-002718-11 (EudraCT Number)
Record Dates: First submitted 2018-09-18; First posted 2018-09-27 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteer
Keywords: Relative Bioavailability and DDI study with MT-7117 and a proton pump inhibitor

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT-7117 BA and DDI (fasted) (Experimental): MT-7117 lower content tablets, higher content tablets, higher content tablets with PPI (fasted), higher content tablets with PPI and acidic beverage (fasted)
  Interventions: Drug: MT-7117; Drug: PPI; Dietary Supplement: Acidic beverage
- MT-7117 food effect and DDI (fed) (Experimental): MT-7117 higher content tablets (fasted and fed), higher content tablets with PPI (fed), higher content tablets with PPI and acidic beverage (fed)
  Interventions: Drug: MT-7117; Drug: PPI; Dietary Supplement: Acidic beverage

INTERVENTIONS:
Drug: MT-7117 — MT-7117
Drug: PPI — Proton pump inhibitor
Dietary Supplement: Acidic beverage — Acidic beverage

SUMMARY:
An open label, multicentre, randomised, 2-cohort, sequential and crossover study to assess the relative oral bioavailability of MT-7117 higher content tablets versus MT-7117 lower content tablets and the pharmacokinetics of MT-7117 under various gastric conditions (fed and fasted, and following administration of a proton pump inhibitor and an acidic beverage) in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* Able to provide written informed consent to participate in this study.
* Healthy and free from clinically significant illness or disease.
* Caucasian male and female subjects aged 18 to 55 years (inclusive) that are willing and able to practice acceptable birth control for the duration of the study, as defined in the Protocol.
* A body weight of ≥50.0 kg and a body mass index (BMI) (Quetelet index) ranging from 18.0 to 30.0 kg/m2 (inclusive) at Screening.
* Subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements.

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Previously having received MT-7117.
* Participation in more than 3 clinical studies* involving administration of an Investigational Medicinal Product (IMP) in the previous year, or any study* involving administration of an IMP within 12 weeks (or, if relevant, 5 half-lives, whichever is the longer) prior to the first dose. (*Disregarding any study Follow-up Periods).
* Subjects who have received any prescribed systemic or topical medication within 14 days (or, if relevant, 5 half-lives; whichever is longer) prior to the first dose of IMP.
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days (or, if relevant, 5 half-lives; whichever is longer) prior to the first dose of IMP.
* Clinically relevant abnormal medical history.
* Family history of long or short QT syndrome, hypokalaemia, syncope or Torsades de Pointes.
* Clinically significant 12-lead electrocardiogram (ECG) abnormalities.
* Blood pressure (supine) at Screening outside the range 90 to 140 mmHg (systolic) or 50 to 90 mmHg (diastolic).
* Presence or history of severe adverse reaction or allergy to any drug.
* Presence or history of drug abuse.
* Presence or history of alcohol abuse.
* Subjects who use tobacco or nicotine-containing products within 3 months.
* Test positive for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV) 1 & HIV 2 antibodies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Pre-dose and up to 48 hours following each single dose
Area under the plasma concentration time curve from time zero to last quantifiable concentration (AUC0-t) | Pre-dose and up to 48 hours following each single dose
Area under the plasma concentration time curve from time zero to infinity (AUC0-inf) | Pre-dose and up to 48 hours following each single dose

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious AEs | up to 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Mitsubishi Tanabe Pharma Europe Ltd
Locations (1):
- Investigational Centre(s), Germany, Germany